CLINICAL TRIAL: NCT06354621
Title: Impact of Vitamin D Supplementation on Fetomaternal Outcomes in Pregnant Females With Latent Tuberculosis Infection: A Randomized Controlled Trial in Lahore-Punjab
Brief Title: Impact of Vitamin D Supplementation on Fetomaternal Outcomes in LTBI Pregnant Females
Acronym: RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, USMAN JAVED IQBAL, Principal Investigator, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: D/185/FIMS
Record Dates: First submitted 2024-03-10; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Maternal and Child Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-A (Control Group) (No Intervention): Participants receiving standard antenatal care without having any vitamin-D supplementation/intervention
- Group-B (2000IU/day) (Experimental): Participants receiving 2000IU/day of Vitamin-D supplementation, in addition to having standard antenatal care
  Interventions: Dietary Supplement: Vitamin-D supplementation
- Group-C (4000IU/day) (Experimental): Participants receiving 4000IU/day of Vitamin-D supplementation, in addition to having standard antenatal care
  Interventions: Dietary Supplement: Vitamin-D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin-D supplementation — Participants receiving a daily dose of vitamin D supplementation
  Arms: Group-B (2000IU/day); Group-C (4000IU/day)

SUMMARY:
The goal of this randomized controlled trial is to see the effect of vitamin D supplementation on fetomaternal outcomes in pregnant females with Latent Tuberculosis infection

The main question[s] it aims to answer are:

If Vitamin D supplementation has any impact on maternal outcomes. If Vitamin D supplementation has any impact on fetal outcomes.

DETAILED DESCRIPTION:
This study aims to see the impact of vitamin D supplementation on fetomaternal outcomes in pregnant females with latent tuberculosis infection. A three-arm (parallel) randomized controlled trial (RCT) will be conducted in a high-burden setting. A calculated sample of 99 (33 in each group) pregnant females with LTBI will be enrolled based on predefined inclusion criteria. Vitamin D supplementation will be given as per study protocols. Group-A (No intervention), Group-B (2000IU/day), Group-C (4000IU/day). To maintain the safety measures throughout the study all the study participants will be monitored for hypervitaminosis D. Informed consent will be obtained from all participants. The study will be conducted after approval by the ethical review board(s). The final analysis will be based on the effect of vitamin D supplementation on pre-defined fetomaternal outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant females aged 18-35 years, already enrolled for delivery in the specified setting coming regularly for prenatal checkups with positive tuberculin skin test

Exclusion Criteria:

* History of active T.B
* Use of any dietary supplement containing more than 400 IU/day (10 mcg/day) of vitamin D within the month before enrolment;
* Presence of any confounders;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 99 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Pre-Eclampsia (Maternal Outcome) | Three months
  Incidence of Pre-eclampsia (percentage of Females having proteinuria on urine dip test with blood pressure > 140/90 mmHg)
Gestational Diabetes Mellitus (Maternal Outcome) | Three months
  Incidence of Gestational diabetes (percentage of females having abnormal glucose intolerance i.e. fasting glucose > 92mg/dL, after using 75g glucose load one-hour glucose > 180mg/dL or two-hour glucose > 153mg/dL)
C/Section delivery (Maternal Outcomes) | Three months
  Incidence of Caesarean delivery (% age of females having surgical delivery of baby via incision on abdomen and uterus)
Low Birth Weight (Foetal Outcome) | One month
  Incidence of low birth weight babies (percentage of neonates weighing <2.5kg)
Pre-Term delivery (Foetal Outcome) | One month
  Incidence of pre-term delivery (percentage of live births before 37 completed gestation weeks)
Apgar Score (Foetal Outcome) | One month
  Apgar scores (The 10-point Apgar score has been used to assess the condition and prognosis of newborn infants throughout the world. Each of five easily identifiable characteristics i.e. heart rate, respiratory effort, muscle tone, reflex irritability, and color is assessed and assigned a value of 0 to 2. The total score is the sum of the five components, and a score of 7 or higher indicates that the baby's condition is good to excellent. The Apgar score is determined at one and five minutes after delivery and is therefore a rapid way to evaluate the physical condition of newborn infants. Of the two scores, the five-minute score has come to be regarded as the better predictor of survival in infancy.)

SECONDARY OUTCOMES:
Improvement in maternal vitamin-D levels | Two-Three months
  To determine whether the baseline vitamin D levels are modified by vitamin D supplementation. (Post intervention mean vitamin-D levels in ng/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Rubeena Zakar, PhD, Study Director — University of the Punjab
Locations (1):
- University of the Punjab, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518